CLINICAL TRIAL: NCT00806130
Title: Health Related Quality of Life and Cognitive Function Among Norwegian Dialysis Patients, a Cross-sectional Study
Brief Title: Health Related Quality of Life and Cognitive Function Among Norwegian Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4.2008.334
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Failure; Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess health related quality of life and its predictors among chronic dialysis patients and to assess cognitive function using 3 different tests.

(undergraduate medical student research project; not published)

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney failure
* Active dialysis treatment
* Aged over 18 years
* Able to read and answer the quality of life questionaire

Exclusion Criteria:

-

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage renal disease and in active dialysis treatment in the Norwegian county of Sør-Trøndelag.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inger Karin Lægreid, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Trondheim, Sør-Trøndelag, Norway